CLINICAL TRIAL: NCT00479154
Title: Pilot Study of Botulinum Toxin Type A for the Treatment of Restless Legs Syndrome
Brief Title: Botulinum Toxin to Treat Restless Legs Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Fatta Nahab, Assistant Clinical Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 070160; 07-N-0160 (Other: Intramural NINDS Protocol # 07-N-0160)
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Results first posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Leg Syndrome; Botulinum Toxin; RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Botulinum Toxins, Type A; onabotulinum toxin A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin A (Experimental): Injection of onabotulinumtoxinA
  Interventions: Drug: Botulinum Toxin A
- Placebo (saline) (Placebo Comparator): Injection of saline placebo
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Drug: Botulinum Toxin A — Maximum dose of 90 units/leg was injected.
  Other Names: onabotulinum toxin

SUMMARY:
This study will test whether botulinum toxin (Botox) may relieve the uncomfortable sensations patients with restless legs syndrome (RLS) experience. RLS is a common movement disorder that causes sensory discomfort and restlessness, most often in the legs, which improves with movement. Although medications are available to treat the disorder, many people experience side effects that prevent them from continuing on the medication. The Food and Drug Administration has approved Botox for other movement disorders and for some cosmetic uses.

People 18 years of age or older with moderate to severe RLS who have been taking RLS medications for more than 6 weeks before entering the study may be eligible to participate. Candidates are screened with a medical history, physical and neurological examinations, blood tests and, for women who can become pregnant, a urine pregnancy test.

Participants are randomly assigned to receive injections of either Botox or placebo (salt water) into up to nine areas of the legs. The correct location of the muscles to be injected is determined by electromyography (EMG), a test that measures the electrical activity of muscles. For surface EMG, electrodes (small metal disks) are filled with a conductive gel and taped to the skin. Needle EMG involves inserting a needle into a muscle. Both methods are used in this study.

At 2 and 4 weeks after the injections, subjects are interviewed by telephone and asked to describe their symptoms, side effects and any improvement they may have noticed. After 12 weeks they return to NIH for injections with the alternate compound; that is, those who received Botox previously are given placebo for the second set of injections, and vice-versa. Subjects are again contacted by telephone 2 and 4 weeks after the injections to report their symptoms, side effects and benefits.

DETAILED DESCRIPTION:
OBJECTIVE:

To evaluate the efficacy of botulinum toxin type A, (BoNT) for the treatment of primary Restless legs syndrome (RLS). We hypothesize that BoNT will be effective at decreasing the deep sensory discomfort of RLS.

STUDY POPULATION:

This protocol is a proof of principle double-blind randomized placebo-BoNT crossover outpatient pilot study of 6 patients diagnosed with moderate to very severe primary RLS.

DESIGN:

All subjects will be evaluated at the NIH Clinical Center by a study investigator to determine eligibility for participation in this protocol. We will obtain a complete medical history, and perform a neurological examination, along with laboratory screening studies. Subjects eligible to participate will receive baseline ratings using the Restless Legs Rating Scale (RLS-RS). Subjects will then be randomized to receive electromyography (EMG)-guided injections of up to 90 units of BoNT or an equivalent volume of saline in each lower extremity, in symptomatic muscles. Subjects will then receive follow up ratings at week 2 and 4 following each injection. Twelve weeks after receiving the first injection, subjects will crossover to receive the alternative compound with similar follow up ratings.

OUTCOME MEASURES:

The primary outcome measure will be mean change from baseline at 4 weeks post-injection on the RLS-RS for placebo and BoNT, while the other pre specified outcomes will evaluate patient reported Clinical Global Impression of Change (CGI-C) scores for each group, duration of effect, and adverse events. Only descriptive statistics will be performed on this limited data sample.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 or older.
* Diagnosed with primary RLS based on presence of a characteristic clinical history and the International restless legs syndrome study group (IRLSSG) diagnostic criteria.
* A minimum score of 11 on the RLS rating scale (this is equivalent to a minimum rating of moderate severity).
* If subjects are on medications for RLS, the medication regimen must be stabilized for greater than 6 weeks prior to entering the study.

EXCLUSION CRITERIA:

* Subjects with any abnormal findings on neurological exam.
* Subjects with a dermatologic disorder that precludes injections in the legs.
* Subjects with a positive urine pregnancy test.
* Subjects without the capacity to give informed consent.
* Subjects taking aminoglycosides, chloroquine, clindamycin, hydroxychloroquine, magnesium sulfate, quinidine, or an anticoagulant.
* Subjects with abnormal clinical chemistry, hematology or urine drug screen by laboratory testing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fatta Nahab, MD, Principal Investigator — NINDS/NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Blasi J, Chapman ER, Link E, Binz T, Yamasaki S, De Camilli P, Sudhof TC, Niemann H, Jahn R. Botulinum neurotoxin A selectively cleaves the synaptic protein SNAP-25. Nature. 1993 Sep 9;365(6442):160-3. doi: 10.1038/365160a0. PMID 8103915

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Botulinum Toxin: Injection into set of leg muscles with Placebo followed by crossover to Botulinum Toxin (90 mU per leg) at week 6.
- Botulinum Toxin Then Placebo: Injection of Botulinum Toxin (90 mU per leg) followed by crossover to placebo at week 6.
Period: Overall Study
Arm/Group | Placebo Then Botulinum Toxin | Botulinum Toxin Then Placebo
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Botulinum Toxin | Botulinum Toxin Then Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.8) | 61.7 (2.5) | 57.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Restless Legs Syndrome Rating Scale
Description: Primary outcome measure will be the mean change from baseline in RLS scale at week 2 following placebo/BTX injections. Scoring criteria are: Mild (score 1-10); Moderate (score 11-20); Severe (score 21-30); Very severe (score 31-40).
Time Frame: Week 2 and Week 4 for each intervention (vs. baseline)
Measure: Mean (Standard Deviation); unit: RLS Rating Score
Groups:
- Placebo: Injection into set of leg muscles with Placebo.
- Botulinum Toxin: Injection of Botulinum Toxin (90 mU per leg).
Arm/Group | Placebo | Botulinum Toxin
Number analyzed (Participants) | 6 | 6
RLS Rating Score
  Week 2 | -5.0 (5.1) | -1.0 (3.5)
  Week 4 | -2.7 (5.9) | -5.0 (6.0)

ADVERSE EVENTS:
Arm/Group | Placebo Then Botulinum Toxin | Botulinum Toxin Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No